CLINICAL TRIAL: NCT00009841
Title: Phase I Trial Of Intratumoral EGFR Antisense DNA And DC-Chol Liposomes In Advanced Oral Squamous Cell Carcinoma
Brief Title: Gene Therapy in Treating Patients With Advanced Head and Neck Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: PCI-98025; CDR0000068414 (Registry Identifier: PDQ (Physician Data Query)); PCI-IRB-980771; NCI-G00-1904
Record Dates: First submitted 2001-02-02; First posted 2004-04-02 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2002-06

CONDITIONS: Head and Neck Cancer
Keywords: untreated metastatic squamous neck cancer with occult primary; recurrent metastatic squamous neck cancer with occult primary; metastatic squamous neck cancer with occult primary squamous cell carcinoma; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the larynx; recurrent squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck

INTERVENTIONS:
Biological: EGFR antisense DNA
Biological: growth factor antagonist therapy
Drug: DC-cholesterol liposome

SUMMARY:
RATIONALE: Gene therapy may kill cancer cells by inhibiting a gene that promotes the development and growth of cancer.

PURPOSE: Phase I trial to study the effectiveness of gene therapy in treating patients who have advanced head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and biological activity of EGFR antisense DNA and DC-chol liposomes in patients with advanced squamous cell carcinoma of the head and neck. II. Determine the toxicity and maximum tolerated dose of this regimen in these patients. III. Determine the antitumor response in patients treated with this regimen. IV. Determine the effect of this regimen on EGFR expression levels, STAT protein expression/activation levels, and apoptosis rates in biopsied tumor cells of these patients.

OUTLINE: This is a dose-escalation study. Patients receive EGFR antisense DNA and DC-chol liposomes intratumorally weekly for 4 weeks. Courses repeat every 4 weeks for up to 6 months in the absence of unacceptable toxicity or disease progression. Cohorts of 3-6 patients receive escalating doses of EGFR antisense DNA and DC-chol liposomes until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 6 patients experience dose-limiting toxicity. Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 20-36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced squamous cell carcinoma of the head and neck Primary or recurrent disease Not amenable to standard therapy (surgery, chemotherapy, or radiotherapy) Second primary lesions allowed Brain metastases allowed after definitive radiotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 8 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL SGOT no greater than 4 times normal Renal: Creatinine no greater than 2 mg/dL Calcium no greater than 10.5 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception (double-barrier method and oral contraception) prior to, during, and for at least 2 weeks after study

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy Surgery: See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 1999-03; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R. Grandis, MD, Study Chair — University of Pittsburgh
Locations (1):
- University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania, United States